CLINICAL TRIAL: NCT01371305
Title: Randomized, Double-Blind, Placebo-Controlled, Multiple Dose, Dose-Escalation Study of STX-100 in Patients With Idiopathic Pulmonary Fibrosis (IPF)
Brief Title: STX-100 in Patients With Idiopathic Pulmonary Fibrosis (IPF)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 203PF201; STX-003 (Other: Stromedix, Inc.)
Record Dates: First submitted 2011-06-03; First posted 2011-06-10 (Estimated); Results first posted 2020-02-28 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Idiopathic Pulmonary Fibrosis (IPF)
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BG00011 (Experimental): Participants will receive 8 consecutive weekly doses of BG00011
  Interventions: Drug: BG00011
- Placebo (Placebo Comparator): Participants will receive 8 consecutive weekly doses of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BG00011 — BG00011 will be administered at varying doses via subcutaneous (SC) injection
  Other Names: STX-100
  Arms: BG00011
Drug: Placebo — Sterile normal saline (0.9% Sodium Chloride for Injection) via Subcutaneous (SC) injections.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of subcutaneously (SC) administered multiple, escalating doses of BG00011 (a humanized monoclonal antibody directed against the alpha v beta 6 (αvβ6) integrin, formerly known as STX-100) in participants with IPF. The Secondary objectives are to estimate the pharmacokinetic (PK) parameters after the 1st dose and after the last dose of multiple, escalating doses of BG00011 in participants with IPF, to assess the immunogenicity of BG00011 in participants with IPF, and to assess the effect of BG00011 on biomarkers isolated from bronchoalveolar lavage (BAL) and peripheral blood in participants with IPF.

DETAILED DESCRIPTION:
This study was previously posted by Stromedix, Inc. In April, 2014, sponsorship of the trial was transferred to Biogen. The study drug name was changed from STX-100 to BG00011 and the study number was changed from STX-003 to 203PF201, to align with sponsor conventions.

ELIGIBILITY:
Key Inclusion Criteria:

1. Clinical features consistent with IPF prior to screening (based on the American Thoracic Society (ATS)/European Respiratory Society (ERS)/Japanese Respiratory Society (JRS)/Latin American Thoracic Association (ALAT) consensus criteria for the diagnosis of IPF).
2. Forced (expiratory) Vital Capacity (FVC) ≥ 50% of predicted value.
3. DLco (corrected for hemoglobin) ≥ 30% predicted value.
4. Oxygen saturation > 90% at rest by pulse oximetry while breathing ambient air or receiving ≤2 L/minute of supplemental oxygen.
5. Residual volume ≤ 120% predicted value.
6. Ratio of Forced Expiratory Volume over 1 second (FEV1) to FVC ≥ 0.65 after the use of a bronchodilator.
7. Other known causes of interstitial lung disease have been excluded (e.g., drug toxicities, environmental exposures, connective tissue diseases).
8. High Resolution Computed Tomography (HRCT) image fulfills the criteria for 'Usual Interstitial Pneumonia (UIP) pattern'.
9. If the HRCT image does not fulfill the criteria for 'UIP pattern' a surgical lung biopsy is necessary for the diagnosis of IPF (lung biopsy performed prior to screening is acceptable). If a lung biopsy has been performed, it must fulfill the histopathological criteria for either 'UIP pattern' or 'probable UIP pattern' with the appropriate HRCT correlate.
10. Adequate bone marrow and liver function.
11. Patient has a life expectancy of at least 12 months.

Key Exclusion Criteria:

1. Findings that are diagnostic of a condition other than UIP on surgical lung biopsy (performed either before or after screening), HRCT imaging, transbronchial lung biopsy, or bronchoalveolar lavage (BAL).
2. Serious local infection or systemic infection within 3 months prior to screening.
3. Treatment with another investigational drug, investigational device, or approved therapy for investigational use within 4 weeks of initial screening.
4. Currently receiving high dose corticosteroid, cytotoxic therapy (e.g., chlorambucil, azathioprine, cyclophosphamide, methotrexate), nintedanib (Ofev®), vasodilator therapy for pulmonary hypertension (e.g., bosentan), unapproved and/or investigational therapy for IPF or administration of such therapeutics within 5 half-lives of the agent prior to initial screening in this study.
5. End-stage fibrotic disease requiring organ transplantation within 6 months

NOTE: Other protocol defined Inclusion/Exclusion Criteria may apply.

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2012-07-16 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (9):
- United States (9):
  - Research Site, San Francisco, California
  - Research Site, Atlanta, Georgia
  - Research Site, Kansas City, Kansas
  - Research Site, Boston, Massachusetts
  - Research Site, Lebanon, New Hampshire
  - Research Site, Cleveland, Ohio
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Nashville, Tennessee
  - Research Site, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The participants were enrolled across 10 sites in the US.
Pre-assignment Details: Forty-one participants were randomized and received at least one dose in the study.
Groups:
- BG00011 0.015 mg: Participants with idiopathic pulmonary fibrosis (IPF) received subcutaneous (SC) injection of 0.015 milligram per kilogram (mg/kg) BG00011 once weekly for 8 doses.
- BG00011 0.1 mg: Participants with IPF received SC injection of 0.1 mg/kg BG00011 once weekly for 8 doses.
- BG00011 0.3 mg: Participants with IPF received SC injection of 0.3 mg/kg BG00011 once weekly for 8 doses.
- BG00011 1.0 mg: Participants with IPF received SC injection of 1.0 mg/kg BG00011 once weekly for 8 doses.
- BG00011 3.0 mg: Participants with IPF received SC injection of 3.0 mg/kg BG00011 once weekly for 8 doses.
- Matching Placebo: Participants with IPF received SC injection of BG00011 matching placebo once weekly for 8 doses.
Period: Overall Study
Arm/Group | BG00011 0.015 mg | BG00011 0.1 mg | BG00011 0.3 mg | BG00011 1.0 mg | BG00011 3.0 mg | Matching Placebo
Started | 6 | 6 | 6 | 7 | 6 | 10
Completed | 6 | 6 | 6 | 5 | 2 | 8
Not Completed | 0 | 0 | 0 | 2 | 4 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 2 | 1 | 0
Not completed — Study terminated by sponsor | 0 | 0 | 0 | 0 | 3 | 1
Not completed — Subject request | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population: The "Safety" population consisted of all participants who received at least one dose of BG00011 or placebo.
Groups:
- Total: Total of all reporting groups
Arm/Group | BG00011 0.015 mg | BG00011 0.1 mg | BG00011 0.3 mg | BG00011 1.0 mg | BG00011 3.0 mg | Matching Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 7 | 6 | 10 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (2.7) | 68 (5.9) | 65 (9.6) | 70 (4.0) | 72 (9.7) | 72 (7.4) | 69 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 1 | 0 | 2 | 1 | 6
  Male | 4 | 6 | 5 | 7 | 4 | 9 | 35
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 6 | 6 | 6 | 7 | 6 | 10 | 41
  Not Hispanic or Latino | 6 | 6 | 6 | 7 | 6 | 10 | 41

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that did not necessarily have a causal relationship with this treatment.
Time Frame: up to Week 19
Population: The "Safety" population consisted of all participants who received at least one dose of BG00011 or placebo.
Measure: Number; unit: Participants
Arm/Group | BG00011 0.015 mg | BG00011 0.1 mg | BG00011 0.3 mg | BG00011 1.0 mg | BG00011 3.0 mg | Matching Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 7 | 6 | 10
Participants | 6 | 5 | 6 | 4 | 6 | 7

2. Secondary Outcome: Time to Reach Maximum Observed Serum Concentration (Tmax) of BG00011
Time Frame: Pre-dose, 8, 24, 48 and 96 hours post-dose on Day 1; pre-dose on Days 8, 15, 22, 29, 36, 43; pre-dose, 24, 48, 96, 168, 336, 504, 672, 1344, 2016 hours post-dose on Day 50
Population: Pharmacokinetic (PK) population = Safety population.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | BG00011 0.015 mg | BG00011 0.1 mg | BG00011 0.3 mg | BG00011 1.0 mg | BG00011 3.0 mg
Number analyzed (Participants) | 6 | 6 | 6 | 7 | 6
hours
  Day 1: number analyzed (Participants) | 2 | 5 | 6 | 7 | 6
  Day 1 | 168 (NA) — Insufficient data to perform analysis. | 101 (42.9) | 132 (39.4) | 134 (60.5) | 96.4 (53.5)
  Day 50: number analyzed (Participants) | 6 | 6 | 6 | 6 | 4
  Day 50 | 42.7 (61.9) | 64.0 (24.8) | 64.0 (51.8) | 32.0 (19.6) | 38.0 (39.4)

3. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of BG00011
Time Frame: as for outcome 2
Population: PK population = Safety population.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | BG00011 0.015 mg | BG00011 0.1 mg | BG00011 0.3 mg | BG00011 1.0 mg | BG00011 3.0 mg
Number analyzed (Participants) | 6 | 6 | 6 | 7 | 6
nanogram per milliliter (ng/mL)
  Day 1: number analyzed (Participants) | 2 | 5 | 6 | 7 | 6
  Day 1 | 71.3 (NA) — Insufficient data to perform analysis. | 335 (178) | 716 (281) | 4370 (1350) | 12900 (3130)
  Day 50: number analyzed (Participants) | 6 | 6 | 6 | 6 | 4
  Day 50 | 134 (44.6) | 1080 (676) | 3170 (1380) | 15400 (5180) | 52800 (17600)

4. Secondary Outcome: Area Under the Serum Concentration Time Curve From Time 0 to Last Quantifiable Observed Concentration AUC(0-t) of BG00011
Time Frame: as for outcome 2
Population: PK population = Safety population.
Measure: Mean (Standard Deviation); unit: hours nanogram per milliliter (hr*ng/mL)
Arm/Group | BG00011 0.015 mg | BG00011 0.1 mg | BG00011 0.3 mg | BG00011 1.0 mg | BG00011 3.0 mg
Number analyzed (Participants) | 6 | 6 | 6 | 7 | 6
hours nanogram per milliliter (hr*ng/mL)
  Day 1: number analyzed (Participants) | 2 | 5 | 6 | 7 | 6
  Day 1 | 9200 (NA) — Insufficient data to perform analysis. | 44800 (24800) | 92600 (40500) | 513000 (264000) | 1730000 (525000)
  Day 50: number analyzed (Participants) | 6 | 6 | 6 | 6 | 4
  Day 50 | 44600 (39400) | 344000 (169000) | 1080000 (554000) | 6370000 (3980000) | 25700000 (17700000)

5. Secondary Outcome: Area Under the Serum Concentration-Time Curve From Time 0 to 168 Hours AUC(0-168) of BG00011
Time Frame: as for outcome 2
Population: PK population = Safety population.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | BG00011 0.015 mg | BG00011 0.1 mg | BG00011 0.3 mg | BG00011 1.0 mg | BG00011 3.0 mg
Number analyzed (Participants) | 6 | 6 | 6 | 7 | 6
hr*ng/mL
  Day 1: number analyzed (Participants) | 2 | 5 | 6 | 6 | 5
  Day 1 | 9200 (NA) — Insufficient data to perform analysis. | 44800 (24800) | 92600 (40500) | 497000 (242000) | 1690000 (438000)
  Day 50: number analyzed (Participants) | 5 | 6 | 6 | 6 | 4
  Day 50 | 21000 (8250) | 159000 (91200) | 465000 (209000) | 2290000 (769000) | 8310000 (2840000)

6. Secondary Outcome: Apparent Terminal Elimination Half Life (T1/2) of BG00011
Time Frame: as for outcome 2
Population: PK population = Safety population. Data for this outcome measure was not collected at Day 1.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | BG00011 0.015 mg | BG00011 0.1 mg | BG00011 0.3 mg | BG00011 1.0 mg | BG00011 3.0 mg
Number analyzed (Participants) | 6 | 6 | 6 | 7 | 6
hour
  Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Day 50: number analyzed (Participants) | 1 | 6 | 6 | 5 | 2
  Day 50 | 178 (NA) — Insufficient data to perform analysis. | 177 (123) | 168 (56.8) | 178 (60.9) | 250 (NA) — Insufficient data to perform analysis.

7. Secondary Outcome: Apparent Terminal Rate Constant [λz]
Time Frame: as for outcome 2
Population: PK population = Safety population. Data for this outcome measure was not collected at Day 1.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | BG00011 0.015 mg | BG00011 0.1 mg | BG00011 0.3 mg | BG00011 1.0 mg | BG00011 3.0 mg
Number analyzed (Participants) | 6 | 6 | 6 | 7 | 6
hour
  Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Day 50: number analyzed (Participants) | 1 | 6 | 6 | 5 | 2
  Day 50 | 0.00390 (NA) — Insufficient data to perform analysis. | 0.00508 (0.00226) | 0.00442 (0.00112) | 0.00423 (0.00123) | 0.00286 (NA) — Insufficient data to perform analysis.

8. Secondary Outcome: Area Under the Concentration Versus Time Curve From Time Zero to Infinity AUC(0-inf) of BG00011
Time Frame: as for outcome 2
Population: PK population = Safety population. Data for this outcome measure was not collected at Day 1.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | BG00011 0.015 mg | BG00011 0.1 mg | BG00011 0.3 mg | BG00011 1.0 mg | BG00011 3.0 mg
Number analyzed (Participants) | 6 | 6 | 6 | 7 | 6
hr*ng/mL
  Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Day 50: number analyzed (Participants) | 1 | 6 | 6 | 5 | 2
  Day 50 | 41900 (NA) — Insufficient data to perform analysis. | 362000 (173000) | 1190000 (690000) | 7250000 (4230000) | 24300000 (NA) — Insufficient data to perform analysis.

9. Secondary Outcome: Apparent Clearance (CL/F) of BG00011
Time Frame: as for outcome 2
Population: PK population = Safety population. Data for this outcome measure was not collected at Day 1.
Measure: Mean (Standard Deviation); unit: milliliter/hour/kilogram (mL/hr/kg)
Arm/Group | BG00011 0.015 mg | BG00011 0.1 mg | BG00011 0.3 mg | BG00011 1.0 mg | BG00011 3.0 mg
Number analyzed (Participants) | 6 | 6 | 6 | 7 | 6
milliliter/hour/kilogram (mL/hr/kg)
  Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Day 50: number analyzed (Participants) | 1 | 6 | 6 | 5 | 2
  Day 50 | 0.913 (NA) — Insufficient data to perform analysis. | 0.758 (0.290) | 0.801 (0.441) | 0.501 (0.172) | 0.486 (NA) — Insufficient data to perform analysis.

10. Secondary Outcome: Apparent Volume of Distribution (Vd/F) of BG00011
Time Frame: as for outcome 2
Population: PK population = safety population. Data for this outcome measure was not analysed on day 1.
Measure: Mean (Standard Deviation); unit: milliliter per kilogram (mL/kg)
Arm/Group | BG00011 0.015 mg | BG00011 0.1 mg | BG00011 0.3 mg | BG00011 1.0 mg | BG00011 3.0 mg
Number analyzed (Participants) | 6 | 6 | 6 | 7 | 6
milliliter per kilogram (mL/kg)
  Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  Day 50: number analyzed (Participants) | 1 | 6 | 6 | 5 | 2
  Day 50 | 234 (NA) — Insufficient data to perform analysis. | 183 (96.0) | 183 (88.0) | 120 (29.8) | 168 (NA) — Insufficient data to perform analysis.

11. Secondary Outcome: Percentage Change (PC) From Baseline in Biomarkers Isolated From Bronchoalveolar Lavage (BAL)
Description: The expression level of 7 genes; Arachidonate 5-lipoxygenase (ALOX5), fibronectin 1 (FN1), Oxidized low density lipoprotein receptor 1 (OLR1), Plasminogen activator inhibitor-1 (PAI-1; aka SERPINE 1), Transglutaminase 2 (TGM2), Triggering receptor expressed on myeloid cells 1 (TREM1), and v-ets erythroblastosis virus E26 oncogene homolog 1 (ETS1) were assessed via BAL as well as a ratio of pSMAD2 to tSMAD2 levels.
Time Frame: Baseline, Day 8 (Follow up)
Population: The "Pharmacodynamic" population consisted of all participants who received at least 1 multiple dose injection of BG00011 and have a corresponding sample collected for BAL and/or blood biomarkers.
Measure: Mean (Standard Deviation); unit: Percentage
Groups:
- Matching Placebo: Participants with IPF received matching placebo.
Arm/Group | BG00011 0.015 mg | BG00011 0.1 mg | BG00011 0.3 mg | BG00011 1.0 mg | BG00011 3.0 mg | Matching Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 7 | 4 | 10
Percentage
  ALOX5; PC at Day 8 (Follow Up): number analyzed (Participants) | 6 | 6 | 6 | 6 | 3 | 9
  ALOX5; PC at Day 8 (Follow Up) | 4.39 (16.560) | -0.25 (11.154) | -5.16 (23.074) | -51.07 (22.942) | -70.90 (14.633) | -7.87 (15.793)
  FN1; PC at Day 8 (Follow Up): number analyzed (Participants) | 6 | 6 | 6 | 6 | 3 | 9
  FN1; PC at Day 8 (Follow Up) | 0.42 (20.776) | -4.83 (22.035) | -16.84 (15.424) | -65.41 (16.174) | -77.42 (17.989) | -8.27 (23.881)
  OLR1; PC at Day 8 (Follow Up): number analyzed (Participants) | 6 | 6 | 6 | 6 | 3 | 9
  OLR1; PC at Day 8 (Follow Up) | -4.79 (31.104) | -1.58 (16.207) | -15.09 (25.235) | -63.64 (18.657) | -77.97 (14.602) | -3.56 (21.215)
  PAI-1; aka SERPINE 1; PC at Day 8 (Follow Up): number analyzed (Participants) | 6 | 6 | 6 | 6 | 3 | 9
  PAI-1; aka SERPINE 1; PC at Day 8 (Follow Up) | 26.98 (55.559) | -28.27 (10.055) | 7.83 (30.064) | -26.06 (38.247) | 71.44 (115.042) | -1.40 (59.537)
  TGM2; PC at Day 8 (Follow Up): number analyzed (Participants) | 6 | 6 | 6 | 6 | 4 | 9
  TGM2; PC at Day 8 (Follow Up) | 0.71 (31.009) | -3.06 (41.757) | -13.17 (35.547) | -53.15 (28.412) | -71.35 (17.449) | 15.06 (59.874)
  TREM1; PC at Day 8 (Follow Up): number analyzed (Participants) | 6 | 6 | 6 | 6 | 3 | 9
  TREM1; PC at Day 8 (Follow Up) | -3.71 (20.135) | -2.01 (16.654) | -7.66 (21.151) | -48.33 (23.511) | -63.13 (13.700) | -12.83 (17.397)
  ETS1; PC at Day 8 (Follow Up): number analyzed (Participants) | 6 | 6 | 6 | 6 | 3 | 9
  ETS1; PC at Day 8 (Follow Up) | 3.16 (53.425) | -11.52 (26.342) | -10.54 (43.866) | 240.59 (245.766) | 103.16 (152.301) | 65.10 (146.690)
  pSMAD2 to tSMAD2; PC at Day 8 (Follow Up): number analyzed (Participants) | 3 | 4 | 5 | 5 | 4 | 7
  pSMAD2 to tSMAD2; PC at Day 8 (Follow Up) | 23.91 (54.293) | -3.33 (29.724) | -39.82 (24.675) | -63.74 (34.674) | -76.20 (14.834) | 28.59 (52.270)

12. Secondary Outcome: Number of Participants With Treatment Emergent Antibodies to BG00011
Time Frame: Up to Week 19
Population: The "Safety" population consisted of all participants who received at least one dose of BG00011 or placebo.
Measure: Number; unit: participants
Arm/Group | BG00011 0.015 mg | BG00011 0.1 mg | BG00011 0.3 mg | BG00011 1.0 mg | BG00011 3.0 mg | Matching Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 7 | 6 | 10
participants | 1 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to Week 19
Description: The "Safety" population consisted of all participants who received at least one dose of BG00011 or placebo.
  The "Other Adverse Events" section includes counts from the "Serious Adverse Events" section.
Arm/Group | BG00011 0.015 mg | BG00011 0.1 mg | BG00011 0.3 mg | BG00011 1.0 mg | BG00011 3.0 mg | Matching Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 1/7 | 0/6 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/6 | 0/6 | 2/7 | 1/6 | 0/10
Other Adverse Events (participants affected / at risk) | 6/6 | 5/6 | 6/6 | 4/7 | 6/6 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BG00011 0.015 mg (N=6) | BG00011 0.1 mg (N=6) | BG00011 0.3 mg (N=6) | BG00011 1.0 mg (N=7) | BG00011 3.0 mg (N=6) | Matching Placebo (N=10)
Atrioventricular Block Complete (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Idiopathic Pulmonary Fibrosis Exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Type II Second-Degree Atrioventricular Block (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Jaw fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BG00011 0.015 mg (N=6) | BG00011 0.1 mg (N=6) | BG00011 0.3 mg (N=6) | BG00011 1.0 mg (N=7) | BG00011 3.0 mg (N=6) | Matching Placebo (N=10)
Injection Site Pain (General disorders) | 0 | 1 | 1 | 0 | 1 | 0
Viral Infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0
Hepatic Enzyme Increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 1 | 1 | 1
Idiopathic Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 3 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Phlebitis Superficial (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 1 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 2 | 0 | 0
Viral Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Upper-Airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Increased Bronchial Secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nasal Discharge Discoloration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Sputum Discolored (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 2 | 0 | 0 | 1
Chest Discomfort (General disorders) | 0 | 1 | 0 | 0 | 1 | 0
Chills (General disorders) | 1 | 0 | 1 | 0 | 0 | 0
Chest Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Infusion Site Bruising (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Injection Site Erythema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Injection Site Paraesthesia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Oedema Peripheral (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vessel Puncture Site Pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 0 | 1 | 0 | 1 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Acute Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Genital Herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 1 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Blood Lactate Dehydrogenase Increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood Pressure Increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Electrocardiogram Qt Prolonged (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Glucose Urine Present (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Oxygen Saturation Decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Protein Urine Present (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Total Lung Capacity Decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Urine Analysis Abnormal (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Urine Leukocyte Esterase Positive (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Cardiac Murmur (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary Function Test Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Muscle Fatigue (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Sensitivity of Teeth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Umbilical Hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 2 | 0 | 0 | 0
Night Sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 0
Bone Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Jaw Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Ligament Sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Limb Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Muscle Strain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Procedural Complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Tooth Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Eye Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Thinking Abnormal (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Angina Pectoris (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Atrioventricular Block Complete (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Atrioventricular Block Second Degree (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Seasonal Allergy (Immune system disorders) | 0 | 3 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Squamous Cell Carcinoma of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Statistical Analysis Plan (2016-05-23): https://cdn.clinicaltrials.gov/large-docs/05/NCT01371305/SAP_000.pdf
  • Study Protocol (2015-07-16): https://cdn.clinicaltrials.gov/large-docs/05/NCT01371305/Prot_001.pdf